CLINICAL TRIAL: NCT06373991
Title: A Phase 1 Study to Evaluate the Safety and Efficacy of ATHENA CAR-T in Subjects With Moderate or Severe Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate the Safety and Efficacy of ATHENA CAR-T in Subjects With Systemic Lupus Erythematosus
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EdiGene Inc. (Industry)
Collaborators: The First Affiliated Hospital of Henan University of Science and Technology (Other); Changping Laboratory (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDI-901-SLE01
Record Dates: First submitted 2024-04-09; First posted 2024-04-18 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-04

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Adult moderate to serve SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — fludarabine; fludarabine phosphate; Injections; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATHENA CAR-T Arm (Experimental): A conditioning chemotherapy regimen will be administered followed by investigational treatment of ATHENA CAR-T
  Interventions: Biological: ATHENA CAR-T; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: ATHENA CAR-T — Phase 1 dose escalation (3+3): dose 1 and dose 2.
  Other Names: ET-901
Drug: Fludarabine — Intravenous injection of fludarabine.
  Other Names: Fludarabine Phosphate for Injection
Drug: Cyclophosphamide — Intravenous injection of cyclophosphamide.
  Other Names: Cyclophosphamide for Injection

SUMMARY:
The goal of this clinical trial is to test ATHENA CAR-T injection in adults with moderate to severe Systemic Lupus Erythematosus. The main question it aims to answer is:

• To evaluate the safety and tolerability of ATHENA CAR-T.

After screening, participants will be subjected to lymphodepletion regimen. After recovery, participants will be injected with ATHENA CAR-T injection and followed up to 24 months.

DETAILED DESCRIPTION:
This study is a single center, one-arm, open label, phase I study aimed at evaluate the safety and effectiveness of ATHENA CAR-T treating moderate to severe SLE patients.

A traditional "3+3" design is used with two doses. DLT is monitored. Safety and effectiveness are followed up until 24 months post infusion of ATHENA CAR-T. Besides safety monitoring, efficacy is evaluated via SLEDAI-2000, BILAG-2004, PGA.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, between 18 and 56 years old;
* diagnosed with SLE according to 2019 EULAR/ACR SLE classifications;
* anti-Nuclear Antigen Ab positive (titer NLT 1:80) and/or dsDNA ab positive and/or Anti-Sm ab positive at screening;
* at screening, SLEDAI-2000 scoring NLT 8 points, if low complement scoring and/or anti-dsDNA ab scoring is available, the SLEDAI-2000 scoring except low complement and anti-dsDNA ab should be NLT 6 points;
* should be subjected to at least 6 months of standard treatment for SLE, and disease active at least two months before screening;
* good organ functions;
* trial participants whose partner is fertile agree to use effective contraceptives til 24 months post transfusion, fertile female participants should have negative urine/blood pregnancy test results (participants who were sterilized or menopause for MT 12 months is not considered fertile);
* voluntary participates this trial and can comprehend and sign ICF.

Exclusion Criteria:

* Had or has active malignancy;
* had been subjected to treatment by CD19 targeted therapy or CAR-T therapy or any gene therapy;
* within 8 weeks before screening, had CNS disease caused by SLE or non-SLE diseases;
* within 8 weeks before screening, had lupus crisis;
* has following kidney diseases: within 8 weeks before randomization, had SLE with serious kidney involvement or need treatment using medications prohibited by protocol to treat active nephritis, or need hemodialysis or need treatment by prednisone MT 100mg/d for longer than 14d or equivalent therapy;
* had serious allergy to any lymphodepletion medication or ingredients of ATHENA CAR-T;
* has uncontrolled fungi, bacterial or viral infection or other infections investigator deemed not suitable to participate in the study;
* combined with other autoimmune disease that needs treatment;
* pregnant or lactating women;
* has other factors that deemed not suitable by investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-07-24 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 0~28 day after treatment
  Dose Limiting Toxicity (DLT) is defined as AEs related to ATHENA CART from infusion till 28 days post infusion.
Frequency of AEs, SAEs, lab abnormalities, AESIs | 0 day to 24 months after treatment
  Monitor grade and frequency of Adverse Events (AEs), Severe Adverse Events (SAEs), abnormal laboratory findings and Adverse Events of Special Interest (AESI).

SECONDARY OUTCOMES:
Efficacy: Percent of patients achieved SRI-4 | 0 to 16 weeks after treatment
  Measure percentage of patients who achieved SRI-4 (Systemic Lupus Erythematosus Responder Index-4) at week 4,8,12,16. SRI-4 response is achieved if SLEDAI-2000 score is lowered NLT 4pt compared to baseline, BILAG-2004 has no new A grade or NMT 1 new B grade, and PGA is not worsen (increase LT 0.3 compare to baseline).
Efficacy: Patients SLEDAI-2000 change compared with baseline | 0 to 16 weeks after treatment
  Compare patients' SLEDAI-2000 (Systemic Lupus Erythematosus Disease Activity Index 2000) value at baseline and week 4,8,12,16. SLEDAI-2000 is an index of range 0 to 105. Higher score indicates stronger disease activity, a score NLT 15 means strong SLE activity.
Efficacy: Patients BILAG-2004 change compared with baseline | 0 to 16 weeks after treatment
  Compare patients' BILAG-2004 (British Isles Lupus Assessment Group index 2004) value at baseline and week 4,8,12,16. Each organ system is graded from A to E, A indicate high disease activity while grade E indicate no disease activity now and then. A is assigned 9 points and E is assigned 0 points.
Efficacy: Percent of patients' PGA not worsen | 0 to 16 weeks after treatment
  Measure percentage of patients whose PGA (Physician Global Assessment) is not worsen (increase LT 0.3 compare to baseline) at week 4,8,12,16. PGA is ranged 0 to 3, score 0 means no disease activity while score 3 means strong disease activity.
Percent of patients responded by BILAG-2004 | 0 to 16 weeks after treatment
  Measure percentage of patients who responded by BILAG-2004 (no new A grade or NMT 1 new B grade) at week 4,8,12,16.
Efficacy: Immunologic parameters | 0 day to 24 months after treatment
  Evaluate the change of immunological parameters. Including of concentration of IgG, IgA, IgM, C3, C4, unit g/L.
Efficacy: Immunologic parameters (cont) | 0 day to 24 months after treatment
  Evaluate the change of immunological parameters. Including concentration of anti-dsDNA antibody, unit IU/ml.

OTHER OUTCOMES:
PK characteristics | 0 day to 24 months after treatment
  Evaluate main PK parameters of ATHENA CAR-T, including Cmax, unit CAR+ T cell/l.
PK characteristics (cont) | 0 day to 24 months after treatment
  Evaluate main PK parameters of ATHENA CAR-T, including Tmax, unit day.
PK characteristics (cont) | 0 day to 24 months after treatment
  Evaluate main PK parameters of ATHENA CAR-T, including AUC0-28d and AUC0-last, both unit are day*CAR+T cell/l.
PD characteristics | 0 day to 24 months after treatment
  Evaluate change of CD19+ cell number, unit CD19 cell/l, before and after infusion of ATHENA CAR-T.
PD characteristics (cont) | 0 day to 24 months after treatment
  Evaluate change of serum cytokine level, including but not limited to TNF-alpha and IFN-gamma, unit pg/ml, before and after infusion of ATHENA CAR-T.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofei Shi, MD, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology
Locations (1):
- The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.